CLINICAL TRIAL: NCT04789746
Title: Ready, Set, Go! A Physical Fitness Intervention for Children With Mobility Challenges
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Chicago Run (Unknown); American Academy of Cerebral Palsy and Developmental Medicine (Other); Spencer Foundation (Unknown)
Responsible Party: Principal Investigator, Theresa Moulton, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00209443
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy; Myelomeningocele; Arthrogryposis; Motor Skills Disorders; Gross Motor Development Delay
MeSH Terms: conditions — Cerebral Palsy; Meningomyelocele; Arthrogryposis; Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Running group (Experimental): Participants that will join the running program.
  Interventions: Behavioral: adapted Chicago Run running program

INTERVENTIONS:
Behavioral: adapted Chicago Run running program — The intervention being piloted is a 6-8 week running program modified from a running curriculum designed for school-aged children. The children will use a RaceRunner device to facilitate their participation, but this device is not explicitly evaluated in this study. Depending on transportation, they may be given access to the device in their home or school between sessions after it has been fit for them. If given access, guardians will be instructed on care and usage.

SUMMARY:
Barriers to keeping and maintaining fitness as a young person with a disability exist across many domains of access to community locations such as fitness centers, so looking outside of these establishments may be necessary to advance fitness. This study is aimed at piloting a program that would address some of these barriers by hosting a modified after school running program with an underserved population in an accessible way. There is a second option to participate outside of school.

ELIGIBILITY:
Inclusion Criteria:

* a medical diagnosis (for example, cerebral palsy) that causes them mobility limitations

Exclusion Criteria:

* concurrent medical condition that would make exercise unsafe,
* are unable to follow simple commands
* have behaviors that would potentially compromise safety of fellow runners or caregivers

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Goal attainment scale | at 8 weeks.
  a tool designed to standardize the setting and scaling of goals in a way that allows for both improvement and regression as a result of intervention.
6 min walk test | baseline
  Participant will walk as far as they can in 6 minutes, as a measure of endurance
6 min walk test | at 8 weeks
  Participant will walk as far as they can in 6 minutes, as a measure of endurance
30 second walk test | baseline
  Participant will walk as fast as they can for 30 seconds, as a measure of speed.
30 second walk test | at 8 weeks
  Participant will walk as fast as they can for 30 seconds, as a measure of speed.
Resting heart rate | baseline
  Participant heart rate after 5 minutes of quiet sitting
Resting heart rate | at 8 weeks
  Participant heart rate after 5 minutes of quiet sitting

SECONDARY OUTCOMES:
Surveys | baseline
  Participants and their parents will answer questions about baseline level of activity, their perception of themselves, and areas of personal strength
Surveys | at 8 weeks
  Participants and their parents will answer questions about baseline level of activity, their perception of themselves, and areas of personal strength
Selective Control Assessment of the Lower Extremity (SCALE) | baseline
  a method of assessing the ability of a participant to isolate motion to an individual joint of the lower extremity. Min score=0; max score=16, a higher score is a better outcome
Selective Control Assessment of the Lower Extremity (SCALE) | at 8 weeks
  a method of assessing the ability of a participant to isolate motion to an individual joint of the lower extremity Min score=0; max score=16, a higher score is a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided